CLINICAL TRIAL: NCT04745975
Title: GUided Treatment Based on Mini-PDX in metastaTIc refractOry Triple Negative Breast Cancer(GUMPTION)：a Prospective Randomized Controlled Single Center Clinical Trial
Brief Title: Guided Treatment Based on Mini-PDX in Metastatic Triple Negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Director of Medical Oncology, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GUMPTION
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Sequence Analysis, RNA; Taxes; eribulin; Vinorelbine; Gemcitabine; Capecitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized treatment guided by Mini-PDX (Experimental): The tumor tissue is used for drug sensitivity test by Mini-PDX, and acquiring the genetic information by RNA-sequence. Patients with mTNBC will receive personalized treatment guided by the experimental results of mini-PDX and RNA sequencing.
  Interventions: Drug: Personalized treatment guided by mini-PDX and RNA sequencing
- Treatment of Physician's Choice (TPC) (Active Comparator): TPC will be administered per standard of care. Patients randomized to TPC will receive chemotherapy, including but not limited to the following agents: nab-paclitaxel, eribulin, vinorelbine, gemcitabine, capecitabine.
  Interventions: Drug: Nab paclitaxel; Drug: Eribulin; Drug: Vinorelbine; Drug: Gemcitabine; Drug: Capecitabine

INTERVENTIONS:
Drug: Personalized treatment guided by mini-PDX and RNA sequencing — Personalized treatment guided by mini-PDX and RNA sequencing
  Arms: Personalized treatment guided by Mini-PDX
Drug: Nab paclitaxel — Nab-paclitaxel 125 mg/m2，ivgtt，d1, 8, 15, q4w
  Arms: Treatment of Physician's Choice (TPC)
Drug: Eribulin — Eribulin 1.4 mg/m2, d1,8 q3w
  Arms: Treatment of Physician's Choice (TPC)
Drug: Vinorelbine — Vinorelbine 25mg/m2 d1,8, q3w
  Arms: Treatment of Physician's Choice (TPC)
Drug: Gemcitabine — Gemcitabine 1000 mg/m2, d1,8, q3w
  Arms: Treatment of Physician's Choice (TPC)
Drug: Capecitabine — Capecitabine 1250 mg/m2 bid po
  Arms: Treatment of Physician's Choice (TPC)

SUMMARY:
Triple-negative breast cancer constitutes 15-20% of cases of breast cancer and is defined by the absence of estrogen receptors, progesterone receptors, and overexpression or gene amplification of HER2. Although the addition of immune checkpoint inhibitors could improve the outcome of patients with metastatic triple-negative breast cancer (mTNBC), chemotherapy has been the standard of care for systemic treatment for patients with mTNBC. Prognoses remain poor, with reported median overall survival estimates of approximately 18 months or less with available treatments. A meta-analysis of seven clinical trials showed that the median objective response rate (ORR) of second or later line of chemotherapy in mTNBC was only 11%.

Patient-derived xenograft (PDX) tumor model, which preserves the histologic and genetic characteristics of patients' tumors, has shown its predictive value of clinical outcomes and are used for preclinical drug evaluation, biomarker identification, biological studies, and personalized medicine strategies. However, long time period and low success rate has limited its application in clinical practice.

Mini patient derived xenograft (miniPDX) offers an effective alternative as it only takes about 7 days for drug sensitivity test and could thus provide guidance for prompt personalized treatment for each patient.

Thus, the investigators conduct this single-center, prospective, randomized controlled clinical study to investigate the efficacy of guided treatment based on Mini-PDX in patients with metastatic refractory triple negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1) Women aged 18-70 years;
* 2) an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* 3) Estimated lifetime is ≥ 3 months;
* 4) Histopathologically confirmed recurrent (unresectable) or metastatic triple-negative breast cancer; ER and PR negative is defined as ER <1% positive, PR <1% positive. HER-2 negative is defined as HER-2 (-) or (1+) by immunohistochemistry, HER-2 (2+) must be tested by FISH with negative result, HER-2 (1+) (1+), FISH is optional and negative;
* 5) Have at least one measurable target lesion according to RECIST 1.1 criteria;
* 6) Biopsy of the tumor lesion and the specimen passes laboratory quality control;
* 7) A minimum of 2 prior cytotoxic chemotherapy regimens (including at least one line of platinum-containing regimen) in metastatic settings are required prior to enrollment in this trial;
* 8) Adequate organ function, i.e. meeting the following criteria.

  1. Hb ≥ 90 g/L (no transfusion within 14 days); ANC ≥ 1.5 × 109 /L; PLT ≥ 75 × 109 /L.
  2. Liver function: total bilirubin TBIL ≤ 1.5×ULN (upper limit of normal); ALT and AST ≤ 3×ULN.
  3. serum Cr ≤ 1.5×ULN.
* 9) Subjects voluntarily joined the study, signed the informed consent form, were compliant and cooperated with the follow-up.

Exclusion Criteria:

* 1）Pregnancy or lactation；
* 2）History of autoimmune disease；
* 3）Anticancer- and radiation therapy-related toxicities have not resolved or downgraded to Grade 1 or less;
* 4) Symptomatic central nervous system (CNS) disease;
* 5) Previous treatment of Immune checkpoint inhibitors;
* 6) History of other malignancies within the past five years, with the exception of cured non-malignant melanoma of the skin and carcinoma in situ of the cervix.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | Through study completion, an expected average of 1 year
  To compare the Objective Response Rate (ORR) of patients who recieve persionalized treatment based on mini-PDX model with ORR of patients who receive Treatment of Physician's Choice (TPC). ORR is defined as the proportion of patients with a confirmed Complete Response (CR) or Partial Response (PR) according to RECIST 1.1. ORR will be calculated based on the Investigator assessment of response. CR = Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm; PR = At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.

SECONDARY OUTCOMES:
Overall Survival | Through study completion, an expected average of 1 year
  Overall survival is defined as the time from the date of randomization to the date of death from any cause. Patients will be followed until their date of death or until final database closure. Patients who are lost-to-follow-up or are alive at the time of analysis will be censored at the time they were last known to be alive or at the date of event cut-off for OS analysis.
Progression-Free Survival | Through study completion, an expected average of 1 year
  Progression-free survival is defined as the time from the date of randomization to the first evidence of documented disease progression as defined by response evaluation criteria in solid tumors (RECIST) v1.1 or death from any cause. Progressive Disease (PD) was at least a 20% increase in the sum of the diameters of target lesions, with reference being the smallest sum on study and an absolute increase of at least 5 mm, or unequivocal progression of non-target lesions, or 1 or more new lesions. If a participant was not known to have died or have objective progression as of the data inclusion cutoff date for the analysis, the PFS time was censored at the last adequate tumor assessment date.
Adverse events | Through study completion, an expected average of 1 year
  Number of participants with adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, M.D., Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No